CLINICAL TRIAL: NCT04357782
Title: Administration of Intravenous Vitamin C in Novel Coronavirus Infection and Decreased Oxygenation (AVoCaDO): A Phase I/II Safety, Tolerability, and Efficacy Clinical Trial
Brief Title: Administration of Intravenous Vitamin C in Novel Coronavirus Infection (COVID-19) and Decreased Oxygenation
Acronym: AVoCaDO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: McGuire Research Institute (Other)
Responsible Party: Principal Investigator, Brian C. Davis, MD, Staff Physician, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Davis 001
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Hypoxia
Keywords: Vitamin C; Ascorbic Acid; Hypoxia; Sepsis; Acute Lung Injury; Acute Respiratory Distress Syndrome; Severe acute respiratory syndrome (SARS)- Coronavirus (CoV)-2
MeSH Terms: conditions — COVID-19; Hypoxia; Sepsis; Acute Lung Injury; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of two or more groups in parallel for the duration of the study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mild hypoxemia (Active Comparator): S/F ratio >250 prior to Vitamin C infusion
  Interventions: Drug: L-ascorbic acid
- Severe Hypoxemia (Active Comparator): S/F ratio ≤250 prior to Vitamin C infusion
  Interventions: Drug: L-ascorbic acid

INTERVENTIONS:
Drug: L-ascorbic acid — 50 mg/kg L-ascorbic acid infusion given every 6 hours for 4 days (16 total doses)
  Other Names: Vitamin C, Ascor

SUMMARY:
Previous research has shown that high dose intravenous vitamin C (HDIVC) may benefit patients with sepsis, acute lung injury (ALI), and the acute respiratory distress syndrome (ARDS). However, it is not known if early administration of HDIVC could prevent progression to ARDS.

We hypothesize that HDIVC is safe and tolerable in Coronavirus disease 2019 (COVID-19) subjects given early or late in the disease course and may reduce the risk of respiratory failure requiring mechanical ventilation and development of ARDS along with reductions in supplemental oxygen demand and inflammatory markers.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability, potential efficacy of high dose intravenous vitamin C (HDIVC) therapy for patients with COVID-19 and decreased oxygenation. COVID-19 is a rapidly evolving pandemic with numerous prediction models suggesting potential shortages in ventilators, ICU beds, and high rates of hospital mortality. Case-series suggest sepsis and the acute respiratory distress syndrome (ARDS) are driving hospitalizations, morbidity (ICU beds, ventilator use, organ failures), and mortality. A therapy is urgently needed to be given early in the disease course in order to attenuate the infectious and inflammatory process, reduce risk of intubation, and reduce progression of organ failure and ARDS. By administering HDIVC at the first objective sign of worsening oxygenation, documented by change in peripheral capillary oxygen saturation (SpO2) to fraction of inspired oxygen (FIO2) ratio (S/F) or decreased SpO2 at baseline (mild hypoxia group), HDIVC may reduce the inflammatory process and development of respiratory failure requiring intubation. We will also enroll patients already in respiratory failure on ventilators (severe hypoxia group) and document safety and tolerability in both cohorts. By calculating ventilator and ICU-free days, we can potentially signal clinically relevant endpoints that could be used in larger trials needed to answer a crucial therapeutic question-can early administration of HDIVC in COVID-19 lead to faster recovery or improve outcomes? Moreover, we will document change in inflammatory markers that are elevated in COVID-19 (d-dimer, C reactive protein (CRP), lactate dehydrogenase (LDH), liver enzymes, and ferritin) to develop a mechanistic understanding and risk stratification of response to HDIVC infusion. Ultimately, if HDIVC is deemed safe and tolerable in hospitalized COVID-19 subjects, a larger clinical trial will be indicated. AVoCaDO will produce safety and tolerability data to test HDIVC in a multi-center, rapid, randomized, placebo-controlled trial of subjects with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with diagnosis of COVID-19 based on positive reverse transcriptase polymerase chain reaction (RT-PCR) SARS-CoV-2 of nasal, oropharyngeal, or bronchoalveolar (BAL) specimen
* Mild deoxygenation defined as S/F ratio decreased by 25% from baseline on admission, or SpO2 <95% breathing ambient air on admission
* Non-childbearing potential or childbearing potential with a negative pregnancy test at screening, and using a reliable method of contraception (i.e., abstinence, hormonal contraception, intrauterine device (IUD), or vasectomized partner)

Exclusion Criteria:

* Known allergy to Vitamin C
* Inability to obtain consent from patient or next of kin
* Chronic kidney disease, stage IV or above (eGFR <30)
* Presence of diabetic ketoacidosis, use of insulin infusion, or frequent need for point-of-care glucose monitoring (>6 times/24 hour period) as determined by treating physician
* History of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Active or history of kidney stone within past 12 months
* Pregnancy
* Enrolled in another COVID-19 clinical trial that does not allow concomitant study drugs

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Davis, MD, Principal Investigator — Staff Physician, GI Division
Locations (1):
- Hunter Holmes Mcguire Veteran Affairs Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowler AA 3rd, Truwit JD, Hite RD, Morris PE, DeWilde C, Priday A, Fisher B, Thacker LR 2nd, Natarajan R, Brophy DF, Sculthorpe R, Nanchal R, Syed A, Sturgill J, Martin GS, Sevransky J, Kashiouris M, Hamman S, Egan KF, Hastings A, Spencer W, Tench S, Mehkri O, Bindas J, Duggal A, Graf J, Zellner S, Yanny L, McPolin C, Hollrith T, Kramer D, Ojielo C, Damm T, Cassity E, Wieliczko A, Halquist M. Effect of Vitamin C Infusion on Organ Failure and Biomarkers of Inflammation and Vascular Injury in Patients With Sepsis and Severe Acute Respiratory Failure: The CITRIS-ALI Randomized Clinical Trial. JAMA. 2019 Oct 1;322(13):1261-1270. doi: 10.1001/jama.2019.11825. PMID 31573637
- [Background] Fowler AA 3rd, Fisher BJ, Kashiouris MG. Vitamin C for Sepsis and Acute Respiratory Failure-Reply. JAMA. 2020 Feb 25;323(8):792-793. doi: 10.1001/jama.2019.21987. No abstract available. PMID 32096845
- [Background] Sindel A, Taylor T, Chesney A, Clark W, Fowler AA 3rd, Toor AA. Hematopoietic stem cell mobilization following PD-1 blockade: Cytokine release syndrome after transplantation managed with ascorbic acid. Eur J Haematol. 2019 Aug;103(2):134-136. doi: 10.1111/ejh.13248. Epub 2019 Jun 7. PMID 31140644
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Background] Fisher BJ, Kraskauskas D, Martin EJ, Farkas D, Puri P, Massey HD, Idowu MO, Brophy DF, Voelkel NF, Fowler AA 3rd, Natarajan R. Attenuation of sepsis-induced organ injury in mice by vitamin C. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):825-39. doi: 10.1177/0148607113497760. Epub 2013 Aug 5. PMID 23917525
- [Background] Fowler Iii AA, Kim C, Lepler L, Malhotra R, Debesa O, Natarajan R, Fisher BJ, Syed A, DeWilde C, Priday A, Kasirajan V. Intravenous vitamin C as adjunctive therapy for enterovirus/rhinovirus induced acute respiratory distress syndrome. World J Crit Care Med. 2017 Feb 4;6(1):85-90. doi: 10.5492/wjccm.v6.i1.85. eCollection 2017 Feb 4. PMID 28224112
- [Background] Kashiouris MG, L'Heureux M, Cable CA, Fisher BJ, Leichtle SW, Fowler AA. The Emerging Role of Vitamin C as a Treatment for Sepsis. Nutrients. 2020 Jan 22;12(2):292. doi: 10.3390/nu12020292. PMID 31978969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 screened upon admission to hospital with positive severe acute respiratory syndrome (SARS)-Coronavirus (CoV)-2 infection and hypoxemia. Seven declined consent, six had history of nephrolithiasis, four had chronic kidney disease stage IV or V, one had glucose-6-phosphate dehydrogenase (G6PD) deficiency.
Period: Overall Study
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Started | 10 | 10
Completed | 9 | 8
Not Completed | 1 | 2
Not completed — Discharged from hospital | 1 | 0
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hypoxemia | Severe Hypoxemia | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 63.5 [40 to 70] | 65.0 [37 to 91] | 63.5 [37 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Admission to Intensive Care Unit (ICU) [Count of Participants; unit: Participants] | 2 | 6 | 8
Hypertension [Count of Participants; unit: Participants] | 6 | 7 | 13
Hyperlipidemia [Count of Participants; unit: Participants] | 5 | 7 | 12
Obesity, any class [Count of Participants; unit: Participants] | 8 | 4 | 12
Diabetes [Count of Participants; unit: Participants] | 2 | 6 | 8
Chronic Obstructive Lung Disease (COPD) [Count of Participants; unit: Participants] | 4 | 2 | 6
Immunocompromised [Count of Participants; unit: Participants] | 4 | 1 | 5
Chronic Kidney Disease (CKD), any stage [Count of Participants; unit: Participants] | 3 | 2 | 5
Chronic liver disease [Count of Participants; unit: Participants] | 2 | 2 | 4
Congestive heart failure [Count of Participants; unit: Participants] | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Related to High Dose Intravenous Vitamin C (HDIVC)
Description: Occurrence of adverse events during study drug infusion as defined in the Ascor package insert ie acute kidney injury (increase in serum creatinine 3x baseline prior to initial HDIVC dose, hemolysis, iatrogenic hypoglycemia, pain at swelling site of infusion, crystalluria on urinalysis (UA) after last HDIVC dose
Time Frame: Days 1-4
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Serious Adverse Reactions
Description: Number of participants with serious adverse events during study drug infusion
Time Frame: Days 1-4
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 10 | 10
Participants | 0 | 2

3. Primary Outcome: Number of Participants With Adverse Reactions
Description: Number of participants with adverse reactions during study drug infusion
Time Frame: Days 1-4
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 10 | 10
Participants | 1 | 2

4. Secondary Outcome: Ventilator-free Days
Description: Documented days free off mechanical ventilation the first 28 days post enrollment
Time Frame: Days 1-28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 10 | 10
days | 28 [0 to 28] | 23.5 [0 to 25]

5. Secondary Outcome: Intensive Care Unit (ICU)-Free Days
Description: Documented days free of ICU admission the first 28 days post enrollment
Time Frame: Days 1-28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 10 | 10
days | 28 [0 to 28] | 13.5 [0 to 22]

6. Secondary Outcome: Hospital-free Days
Description: Documented days free of hospital admission the first 28 days post enrollment
Time Frame: Days 1-28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 10 | 10
days | 21.5 [21 to 28] | 8.5 [5 to 24]

7. Secondary Outcome: All-cause Mortality
Description: Incidence of mortality at 28 days by all causes
Time Frame: Days 1-28
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 10 | 10
Participants | 0 | 3

8. Secondary Outcome: Change in S/F Ratio During High Dose Intravenous Vitamin C (HDIVC)
Description: oxygen saturation by pulse oximetry (SpO2) will be divided by fraction of inspired oxygen (FiO2) at start of study infusion and compared with S/F ratio at end of study infusion
Time Frame: Days 1-4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 10 | 10
ratio | 108 (121) | 26 (140)

9. Secondary Outcome: C-reactive Protein (CRP)
Description: The difference in serum CRP during HDIVC infusion reported in mg/dL
  Local lab with upper measurement limit of 19 mg/dL
  The change was determined from two time points ie Day 4value minus Day 1 value.
Time Frame: Days 1-4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 9 | 9
mg/dL | -3.8 (5.1) | -2.0 (6.7)

10. Secondary Outcome: Lactate Dehydrogenase (LDH)
Description: The difference in LDH during HDIVC infusion will be reported in IU/L
  The change was determined from two time points ie Day 4 value minus Day 1 value.
Time Frame: Days 1-4
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 9 | 8
IU/L | -42 (131) | 118 (497)

11. Secondary Outcome: D-dimer
Description: The difference in D-dimer during HDIVC infusion will be reported in ug/mL
  The change was determined from two time points ie Day 4 value minus Day 1 value.
Time Frame: Days 1-4
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 8 | 9
ug/mL | -0.21 (0.72) | 3.71 (6.9)

12. Secondary Outcome: Lymphocyte Count
Description: The difference in lymphocyte count during HDIVC infusion will be reported in 10^3 cells/uL
  The change was determined from two time points ie Day 4 value minus Day 1 value.
Time Frame: Days 1-4
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 8 | 7
10^3 cells/uL | 329 (514) | 276 (581)

13. Secondary Outcome: Neutrophil to Lymphocyte Ratio (NLR)
Description: The NLR will be calculated by dividing the absolute neutrophil count (10e3/uL) over the absolute lymphocyte count (10e3/uL)
  The change was determined from two time points ie Day 4 value minus Day 1 value.
Time Frame: Days 1-4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 8 | 7
ratio | -0.89 (4.8) | -0.04 (5.0)

14. Secondary Outcome: Serum Ferritin
Description: The difference in serum ferritin will be calculated from the start of HDIVC infusion to day 4 and reported as ng/mL
  The change was determined from two time points ie Day 4 value minus Day 1 value.
Time Frame: Days 1-4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
Number analyzed (Participants) | 9 | 8
ng/mL | -299 (449) | -1170 (2997)

ADVERSE EVENTS:
Time Frame: Data were collected systemically daily during study drug infusion and by electronic record review over the course of 28 days since study enrollment
Arm/Group | Mild Hypoxemia | Severe Hypoxemia
All-Cause Mortality (participants affected / at risk) | 0/10 | 3/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 3/10
Other Adverse Events (participants affected / at risk) | 5/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hypoxemia (N=10) | Severe Hypoxemia (N=10)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Mechanical intubation due to worsening acute hypoxemic respiratory failure due to COVID-19.
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) — Acute kidney injury, stage 3 due to ischemia
Pulseless Electrical Activity Arrest (Cardiac disorders) | 0 (0) | 2 (2) — Pulse-less electrical activity arrest from acute hypoxemic respiratory failure due to COVID-19, day 2
ischemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Hepatic Failure/ischemic hepatitis post pulseless electrical activity arrest
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hypoxemia (N=10) | Severe Hypoxemia (N=10)
Elevated ALT (Hepatobiliary disorders) | 0 (0) | 1 (1) — Elevated ALT/DILI with peak ALT of 423 IU/L, likely due to tocilizumab
Nausea, self-limited (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) — Deep vein thrombosis left posterior tibial
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — +methicillin-resistant Staphylococcus aureus (MRSA) sputum culture
Bacteremia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — coagulase-negative
Chest Pain (General disorders) | 1 (1) | 2 (2) — Mild, self limited
Elevated ALT (Hepatobiliary disorders) | 0 (0) | 1 (1) — likely related to remdesivir, resolved
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — < 4 episodes per day
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04357782/Prot_SAP_000.pdf